CLINICAL TRIAL: NCT04786665
Title: Impact of Strawberries on Cognition, and Vascular and Cardiometabolic Markers in Older Healthy Adults
Brief Title: Strawberries, Cognition, and Vascular Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Shirin Hooshmand, Professor, San Diego State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 59650A
Record Dates: First submitted 2021-03-03; First posted 2021-03-08 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Aging; Healthy Aging
Keywords: Cognition; Motor control; Vascular health

STUDY DESIGN:
Intervention Model Description: Using a randomized crossover study design, the effects will be compared to the effects of 8 wk intake of a placebo drink-mix (with a 4 wk wash-out period between trials).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strawberry powder (Experimental): Participants consume 1 package of standard strawberry powder (26 g) daily for 8 weeks
  Interventions: Other: Strawberry
- Placebo group (Placebo Comparator): Participants consume 1 package of placebo powder (26 g) daily for 8 weeks
  Interventions: Other: Placebo group

INTERVENTIONS:
Other: Strawberry — Freeze dried strawberry powder
  Arms: Strawberry powder
Other: Placebo group — Comparative placebo powder
  Arms: Placebo group

SUMMARY:
The primary objective of this study is to investigate the effects of strawberries on cognitive responses, motor control function, and vascular and cardiometabolic risk markers in healthy older adults.

DETAILED DESCRIPTION:
To achieve the objectives, 40 healthy men and women ≥65 years of age will consume 26 g of freeze-dried strawberries in the form of a drink-mix daily for 8 wk. Using a randomized crossover study design, the effects will be compared to the effects of 8 wk intake of a placebo drink-mix (with a 4 wk wash-out period between trials). Cognitive function measurements will be performed at baseline and 8 wk. Additionally, at each timepoint, flow-mediated vasodilation and blood pressure will be measured followed by collection of fasting blood samples to assess glucose, insulin, blood lipids (free fatty acids, triacylglycerol, total cholesterol, LDL cholesterol, and HDL cholesterol), inflammatory markers (interleukins 6 and 18), and markers of oxidative stress (oxidized LDL-C and malondialdehyde).

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women 65 years and older

Exclusion Criteria:

* stroke or myocardial infarction
* neurological disorders:
* epilepsy,
* multiple sclerosis,
* Parkinson's disease,
* stroke
* known metabolic disorders:
* liver,
* renal
* clinically diagnosed diabetes
* drug treatment for lipid reduction or hypertension,
* psychiatric medication use

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in processing speed (cognition) at 8 weeks | At baseline, at 8 weeks
  using Pattern Comparison Processing Speed Test
Change from baseline in executive function (cognition) at 8 weeks | At baseline, at 8 weeks
  using Dimensional Change Card Sort Test; Flanker Inhibitory Control and Attention Test
Change from baseline in working memory (cognition) at 8 weeks | At baseline, at 8 weeks
  using List Sorting Working Memory Test
Change from baseline in episodic memory (cognition) at 8 weeks | At baseline, at 8 weeks
  using Picture Sequence Memory Test
Change from baseline in working memory (cognition) at 8 weeks | At baseline, at 8 weeks
  using Picture Vocabulary Test; Oral Reading Recognition Test

SECONDARY OUTCOMES:
Change from baseline in Vascular health at 8 weeks | At baseline, at 8 weeks
  to better understand how changes in the gut microbiota through fruit consumption are linked to changes in health outcomes, we will assess endothelial function via flow-mediated vasodilation and risk factors for cardiometabolic dysfunction in fasting blood samples collected at baseline and after 8 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Shirin Hooshmand, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Delaney K, Tsang M, Kern M, Rayo VU, Jason N, Hong MY, Liu C, Hooshmand S. Strawberries modestly improve cognition and cardiovascular health in older adults. Nutr Metab Cardiovasc Dis. 2025 Aug;35(8):104018. doi: 10.1016/j.numecd.2025.104018. Epub 2025 Mar 18. PMID 40199714